CLINICAL TRIAL: NCT06976320
Title: Deep Rectus Sheath Block for Postoperative Analgesia in Patients Undergoing Laparoscopic Cholecystectomy
Brief Title: Deep Rectus Sheath Block for Laparoscopic Cholecystectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Anestezi4
Record Dates: First submitted 2025-05-09; First posted 2025-05-16 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Cholecystectomy, Laparoscopic; Anesthesia; Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): The patients in Control Group will be received patient controlled analgesia with morphine for postoperative analgesia
  Interventions: Other: Intravenous morphine patient control analgesia
- Deep rectus sheath block group (Active Comparator): The patients in deep rectus sheath block group will be received deep rectus sheath block and patient controlled analgesia with morphine for postoperative analgesia
  Interventions: Other: Intravenous patient control analgesia; Other: Deep rectus sheath block

INTERVENTIONS:
Other: Intravenous morphine patient control analgesia — 24-hour morphine consumption will be recorded
  Arms: Control group
Other: Intravenous patient control analgesia — 24-hour morphine consumption will be recorded
  Arms: Deep rectus sheath block group
Other: Deep rectus sheath block — Deep rectus sheath block will be administered at the end of the surgery.
  Arms: Deep rectus sheath block group

SUMMARY:
Postoperative pain after laparoscopic cholecystectomy can be considerable. Regional techniques such as erector spinae plane (ESP) block or transversus abdominis plane (TAP) block may be suitable for patients at increased risk of postoperative pain. The deep rectus sheath block is a novel block which is a modified version of the conventional rectus sheath block. It was reported in a few case reports that, it may be used for postoperative analgesia in patients undergoing laparoscopic cholecystectomy. The aim of this study is to investigate the postoperative analgesic efficacy of deep rectus sheath block in patients undergoing laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
Patients scheduled for elective laparoscopic gastrectomy will be separated into 2 groups: Control Group and Deep Rectus Sheath Block Group. Patients in Control Group will be received patient controlled analgesia with morphine for postoperative analgesia. Patients in Deep Rectus Sheath Block Group will be performed Deep Rectus Sheath Block at the end of the surgery, along with patient controlled analgesia with morphine for postoperative analgesia. Morphine consumption for first postoperative 24 hours, numerical rating scale scores, amount of rescue analgesic drug, incidence of postoperative nausea and vomiting will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years
* Patients with American Society of Anesthesiology (ASA) physical status I-II
* Patients scheduled for a laparoscopic cholecystectomy

Exclusion Criteria:

* Allergy to local anesthetics
* Coagulopathy
* Skin infection at the deep rectus sheath block area
* Advanced hepatic or renal failure
* Chronic pain syndromes
* Alcohol or drug abuse
* Severe pulmonary and/or cardiovascular disease
* Psychiatric disorders

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-09 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Morphine consumption | Postoperative 24 hours
  The amount of morphine required by the patient and given by the device will be recorded for the first 24 hours.

SECONDARY OUTCOMES:
Postoperative numerical rating scale scores | Postoperative 24 hours
  Postoperative pain will be assessed using a numerical rating scale (NRS) (from 0 = no pain to 10 = maximum possible pain) for the first 24 hours.
Rescue analgesic drug requirement | Postoperative 24 hours
  The amount of rescue analgesic in mg required by the patient will be recorded for the first 24 hours.
Incidence of postoperative nausea and vomiting | Postoperative 24 hours
  Number of patients developing postoperative nausea and vomiting will be recorded for the first 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Taylan Sahin, M.D., Principal Investigator — Istinye University; Ali Sait Kavakli, M.D., Principal Investigator — Istinye University
Locations (1):
- Istinye University Hospital, Istanbul, Turkey (Türkiye)